CLINICAL TRIAL: NCT03732248
Title: Altering Memories That Increase Risk of Relapse in Alcohol Use Disorders: A Translational Clinical Neuroscience Pilot Investigation of a Novel Pharmacological Agent
Brief Title: Altering Memories That Increase Risk of Relapse in Alcohol Use Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00073523
Record Dates: First submitted 2018-11-01; First posted 2018-11-06 (Actual); Results first posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Alcohol Use Disorder; Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — Sirolimus; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rapamycin (sirolimus) 15mg (Active Comparator): Rapamycin (sirolimus) is administered in three 5mg oral capsules. This administration happens once during the first visit.
  Interventions: Drug: Rapamycin
- Placebo (Placebo Comparator): Placebo is administered in three 5mg oral capsules. This administration happens once during the first visit.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rapamycin — Immunosuppressive drug
  Other Names: Sirolimus
  Arms: Rapamycin (sirolimus) 15mg
Drug: Placebo — Inert drug
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the effects of rapamycin (sirolimus) versus a placebo, an inactive substance, on responses to alcohol cues in individuals with alcohol use disorder. Rapamycin (sirolimus) is a FDA-approved antibiotic and immunosuppressive drug that is currently used to (a) prevent organ transplant recipients from rejecting their transplants (b) treat cardiovascular diseases, and (c) treat some forms of cancer. Rapamycin (sirolimus) is not FDA-approved to treat alcohol use disorder. The use of rapamycin (sirolimus) in this study is investigational, meaning that the study medication is not a proven treatment for alcohol use disorder. The study will examine the medication's use as a potential treatment for alcohol use disorder, as well as how safe and tolerable it is to take.

ELIGIBILITY:
Inclusion Criteria:

* Must be treatment-seekers
* Meet criteria for alcohol use disorder
* Must be able to provide informed consent and function at an intellectual level sufficient to allow accurate completion of all assessment instruments
* Must use one of the following methods of birth control: oral contraceptives, barrier methods (diaphragm or condoms with spermicide or both), surgical sterilization, use of an intra-uterine contraceptive device, or complete abstinence from sexual intercourse
* Must live within a 50-mile radius of our research program and have reliable transportation,
* Must consent to remain abstinent from alcohol and all non-prescription drugs prior to medication administration and testing sessions
* Must consent to fast for a two-hour period prior to medication administration
* Must consent to random assignment to the rapamycin vs. placebo conditions.

Exclusion Criteria:

* Cannot be undergoing other alcohol cessation treatment
* Cannot be pregnant, nursing, or of childbearing potential and not using birth control
* Cannot have evidence of or a history of significant endocrine, cardiovascular, pulmonary, renal, or neurological disease
* Cannot have significant liver impairment
* Cannot have an existing infection or immune system disorder
* Cannot have a history of or current psychotic disorder, severe major depression, or bipolar affective disorder
* Cannot currently take anti-arrythmic agents, psychostimulants, or any other agents known to interfere with heart rate and skin conductance monitoring
* Cannot have known or suspected hypersensitivity to macrolide compounds (such as rapamycin/sirolimus)
* Cannot currently take medications that could adversely interact with the study medication, including but not limited to significant inhibitors of CYP2D6 or CYP3A4 (voriconazole, fluconazole, itraconazole, erythromycin, clarithromycin, diltiazem, verapamil, etc.), or significant inducers of CYP3A4, such as anticonvulsants (carbamazepine, phenobarbital, phenytoin, etc.) and antibiotics (rifabutin, rifapentine, etc.)
* Cannot have a history of thrombocytopenia, idiopathic thrombocytopenia purpura (ITP) or have a platelet count of less than 100,000 cells per mm3
* Cannot have any unhealed wounds
* Cannot have any planned surgeries within the next month, including surgical dental procedures
* Cannot have a history of complicated alcohol withdrawal symptoms (including, but not limited to, symptoms such as seizures, hallucinations, and high blood pressure)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Saladin, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rapamycin (Sirolimus) 15mg | Placebo
Started | 11 | 10
Completed | 10 | 10
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rapamycin (Sirolimus) 15mg | Placebo | Total
Number analyzed (Participants) | 11 | 10 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.1 (9.9) | 37.8 (7.8) | 40.6 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 12
  Male | 4 | 5 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 10 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 10 | 21

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Safety of a Single 15 mg Dose of Rapamycin (Sirolimus) at First Visit.
Description: Safety will be monitored through adverse events checks by the study physician assistant (PA). The study PA will use the Monitoring of Side-Effects Scale (MOSES) to track if there are any adverse effects. Participants will be recorded as those who report any adverse event vs. no adverse events.
Time Frame: MOSES will be assessed at the first study visit on day 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Rapamycin (Sirolimus) 15mg | Placebo
Number analyzed (Participants) | 11 | 10
Participants | 0 | 3

2. Primary Outcome: Evaluate Safety of Rapamycin (Sirolimus) at Second Visit.
Description: as for outcome 1
Time Frame: MOSES will be assessed at the second study visit, 24 hours after medication administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Rapamycin (Sirolimus) 15mg | Placebo
Number analyzed (Participants) | 10 | 10
Participants | 2 | 6

3. Primary Outcome: Evaluate Safety of Rapamycin (Sirolimus) at Third (Last) Visit.
Description: as for outcome 1
Time Frame: MOSES will be assessed at the third study visit, approximately 10 days after medication administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Rapamycin (Sirolimus) 15mg | Placebo
Number analyzed (Participants) | 10 | 10
Participants | 3 | 0

4. Secondary Outcome: Drinking Days Between Visit 2 and Visit 3
Description: Participants will be given a timeline to record any drinking that occurs between visits 2 and 3.
  Time line follow back procedures were used to record daily drinking behavior for all study days; recorded as standard drinks. The total number of days where drinking was recorded is summed for each participants during the study window.
Time Frame: At participant's last study visit, approximately 10-14 days.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Rapamycin (Sirolimus) 15mg | Placebo
Number analyzed (Participants) | 10 | 10
Days | 10.5 [4 to 12] | 8 [5 to 10]

5. Secondary Outcome: Drinks Per Drinking Day Between Visit 2 and Visit 3
Description: Participants will be given a timeline to record any drinking that occurs between visits 2 and 3.
  Time line follow back procedures were used to record daily drinking behavior for all study days; recorded as standard drinks.
Time Frame: At participant's last study visit, approximately 10 days.
Measure: Mean (Standard Deviation); unit: Standard Drinks/day
Arm/Group | Rapamycin (Sirolimus) 15mg | Placebo
Number analyzed (Participants) | 10 | 10
Standard Drinks/day | 4.8 (1.5) | 3.2 (2.2)

6. Secondary Outcome: Heavy Drinking Days Between Visit 2 and Visit 3
Description: Participants will be given a timeline to record any drinking that occurs between visits 2 and 3.
  Time line follow back procedures were used to record daily drinking behavior for all study days; recorded as standard drinks. Heavy drinking days are defined as >=5 drinks per day for Males and >=4 drinks per day for Females.
Time Frame: At participant's last study visit, approximately 10 days.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Rapamycin (Sirolimus) 15mg | Placebo
Number analyzed (Participants) | 10 | 10
Days | 5 [2 to 11] | 2 [2 to 4]

ADVERSE EVENTS:
Time Frame: Participants were assessed for adverse events between baseline and follow-up for a total of three weeks.
Arm/Group | Rapamycin (Sirolimus) 15mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 0/11 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-29): https://cdn.clinicaltrials.gov/large-docs/48/NCT03732248/Prot_SAP_000.pdf